CLINICAL TRIAL: NCT02320396
Title: A Phase III, Multi-Center, Randomized, Placebo-Controlled, Double-Blind Trial to Study the Efficacy and Safety of MK-4117 in Japanese Subjects With Seasonal Allergic Rhinitis
Brief Title: Efficacy and Safety Study of Desloratadine (MK-4117) in Japanese Participants With Seasonal Allergic Rhinitis (MK-4117-204)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4117-204; 152861 (Registry Identifier: JAPIC-CTI); MK-4117-204 (Other: Merck Registration Number)
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desloratadine (Experimental): After a 1-week single-blinded placebo run-in during which SAR symptoms are confirmed (Confirmation of Symptom Period), participants receive double-blinded desloratadine (one 5 mg tablet) orally (PO) once daily (QD) in the morning for 2 weeks during the Treatment Period.
  Interventions: Drug: Desloratadine 5 mg
- Placebo (Placebo Comparator): After a 1-week single-blinded placebo run-in during which SAR symptoms are confirmed (Confirmation of Symptom Period), participants receive double-blinded placebo (one tablet) PO QD in the morning for 2 weeks during the Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desloratadine 5 mg — Desloratadine 5 mg tablets
  Arms: Desloratadine
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This is an efficacy and safety study of desloratadine (MK-4117) in Japanese participants with seasonal allergic rhinitis (SAR). The primary hypothesis of this study is that the change from Baseline in Total Nasal Symptom Score (TNSS) is improved by desloratadine compared to placebo.

DETAILED DESCRIPTION:
This study consists of a one-week Symptom Confirmation Period during which participants undergo a single-blinded placebo run-in, a two-week double-blind Treatment Period and a two-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Has at least a 2-year history of seasonal allergic rhinitis with typical symptoms
* Male or female who is unlikely to conceive: a surgically sterilized female, female who has reached natural menopause, or is of reproductive potential and agrees to either remain abstinent or use (or have her partner use) 2 acceptable methods of birth control from study start through 14 days after the last dose of study drug.

Exclusion Criteria:

* Has a lower respiratory tract infection or has a nasopharyngolaryngeal infection (acute upper respiratory tract infection, acute pharyngolaryngitis, or acute tonsillitis, etc.) requiring treatment
* Has a coexisting infection or systemic mycosis for which there are no effective antibiotics
* Has asthma that is under treatment and/or uncontrolled
* Has nasal septum ulcers, nasal surgery, or nasal trauma which have not healed
* Has vasomotor rhinitis or eosinophilic rhinitis
* Has a history of hypersensitivity to antihistamines or ingredients of study drug
* Has had treatment with corticosteroids (oral, injectable, suppository, depot drugs [injectable]) or immunological drugs within 28 days prior to Visit 2
* Is currently receiving treatment with another investigational drug or has received an investigational drug within prior 3 months
* Has started specific desensitization therapy (allergen immunotherapy) or nonspecific allassotherapy (Histaglobin, vaccine therapy, etc.) or who has received such therapies within prior 3 months
* Has received coagulation or resection using laser therapy etc. for treatment for nasal symptoms
* Will receive nasal nebulizer therapy and/or thermotherapy during study period
* Has severe hepatic, renal, cardiac, hematological disease, or other serious coexisting diseases and whose general condition is poor
* Has a history of malignancy or clinically important hematological disorder, except for adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix
* Has a history of severe drug allergy (e.g. anaphylactoid reaction)
* Is pregnant or lactating or may be pregnant
* Is planning a remote trip for more than 1 day during the Symptom Confirmation Period or for more than 2 days during the Treatment Period.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okubo K, Maeda Y, Oshima N, Hisada S. A Phase III clinical trial of desloratadine in Japanese subjects with seasonal allergic rhinitis: A randomized controlled trial. Arerugi. 2016;32(11):863-876.. [in Japanese] https://mol.medicalonline.jp/archive/search?jo=an9cltmd&ye=2016&vo=32&issue=11

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with seasonal allergic rhinitis (SAR) were recruited at 3 study sites in Japan.
Pre-assignment Details: Of 1148 participants screened, 449 were enrolled in the study and randomized to oral (PO) once daily (QD) Desloratadine (n=224) or Placebo (n=225). One participant randomized to Desloratadine was not treated due to withdrawn consent.
Groups:
- Desloratadine: After a 1-week single-blinded placebo run-in during which SAR symptoms are confirmed (Confirmation of Symptom Period), participants receive double-blinded desloratadine (one 5 mg tablet) PO QD in the morning for 2 weeks during the Treatment Period.
Period: Overall Study
Arm/Group | Desloratadine | Placebo
Started | 224 | 225
Treated (Full Analysis Set) | 223 | 225
Completed | 220 | 221
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Desloratadine | Placebo | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (10.9) | 39.8 (10.9) | 39.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 131 | 261
  Male | 94 | 94 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) During 2 Weeks of Therapy
Description: The TNSS was used to evaluate participant nasal symptoms of: sneezing (daily frequency of attacks scored from 0 [<1 time or "none"] to 4 [≥21 times]), rhinorrhea (daily frequency of blowing nose scored from 0 [<1 time or "none"] to 4 [≥21 times]), nasal congestion (scored from 0 [no nasal blockage] to 4 [completely obstructed all day]), and nasal itching (scored from 0 [none] to 4 [nose is itchy, requiring frequent rubbing or blowing nose) as rated in the participant's diary. The TNSS was the sum of the 4 nasal symptom sub-scores. TNSS scores ranged from 0 to 16, with a higher score indicating more frequent/severe nasal symptoms. Baseline (BL) measurement was an average of scores for 3 days prior to treatment (during Confirmation of Symptom Period). Post-BL measurement was an average from Day 1 to Day 13 (2 week average). Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to Day 13 (Weeks 1 through 2 average) of double-blind treatment
Population: The Full Analysis Set (FAS); all randomized participants who took ≥1 dose of study treatment, and have a BL (average of score for 3 days prior to treatment) observation or one post BL observation (average score of 2 weeks).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale | -1.41 [-1.64 to -1.19] | -0.59 [-0.81 to -0.36]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; The LS mean change from BL to post BL (average score of 2 weeks) in TNSS was estimated using a constrained longitudinal data analysis (cLDA) model, where both BL and post-BL measurements (average score of 2 weeks) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in Least Squares (LS) Means = -0.83, 95% CI 2-sided [-1.14 to -0.51]

2. Primary Outcome: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an AE.
Time Frame: Up to 4 weeks (Up to 2 weeks after last dose of study drug)
Population: All Participants as Treated (APaT); all participants who received ≥1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
participants | 19 | 13

3. Primary Outcome: Number of Participants Who Discontinue Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 2 weeks
Population: APaT; all participants who received ≥1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
participants | 2 | 2

4. Secondary Outcome: Change From Baseline in TNSS for Week 1 and Week 2 of Double-blind Treatment
Description: The TNSS was used to evaluate participant nasal symptoms of: sneezing (daily frequency of attacks scored from 0 [<1 time or "none"] to 4 [≥21 times]), rhinorrhea (daily frequency of blowing nose scored from 0 [<1 time or "none"] to 4 [≥21 times]), nasal congestion (scored from 0 [no nasal blockage] to 4 [completely obstructed all day]), and nasal itching (scored from 0 [none] to 4 [nose is itchy, requiring frequent rubbing or blowing nose) as rated in the participant's diary. The TNSS was the sum of the 4 nasal symptom sub-scores. TNSS scores ranged from 0 to 16, with a higher score indicating more frequent/severe nasal symptoms. Baseline (BL) measurement was an average of scores for 3 days prior to treatment (during Confirmation of Symptom Period). Post-BL measurement for Week 1 was an average from Day 1 to Day 7 and post-BL measurement for Week 2 was an average from Day 8 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to 7 (Week 1 average), Day 8 to 13 (Week 2 average) of double-blind treatment
Population: The FAS; all randomized participants who took ≥1 dose of study treatment, and have a BL (average of score for 3 days prior to treatment) observation or one post BL observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Week 1 | -1.19 [-1.42 to -0.96] | -0.38 [-0.61 to -0.15]
  Week 2 | -1.69 [-1.96 to -1.41] | -0.84 [-1.12 to -0.57]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL in TNSS at Week 1: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in TNSS was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.82, 95% CI 2-sided [-1.14 to -0.50]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL in TNSS at Week 2: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in TNSS was estimated using a cLDA model, where both BL and post- BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.84, 95% CI 2-sided [-1.23 to -0.46]

5. Secondary Outcome: Change From Baseline to Week 1 in Each Nasal Symptom Sub-Score (Sneezing, Rhinorrhea, Nasal Congestion and Nasal Itching)
Description: Nasal symptoms sub-scores rated in the participant's diary included sneezing (daily frequency of attacks scored from 0 [<1 time or "none"] to 4 [≥21 times]), rhinorrhea (daily frequency of blowing nose scored from 0 [<1 time or "none"] to 4 [≥21 times]), nasal congestion (scored from 0 [no nasal blockage] to 4 [completely obstructed all day]), and nasal itching (scored from 0 [none] to 4 [nose is itchy, requiring frequent rubbing or blowing nose). Nasal symptom sub-scores ranged from 0 to 4, with a higher score indicating more frequent/severe nasal symptoms. BL measurement was an average of scores for 3 days prior to treatment (during Confirmation of Symptom Period). Post-BL measurement for Week 1 was an average of scores from Day 1 to Day 7. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to 7 (Week 1 average) of double-blind treatment
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Sneezing | -0.39 [-0.47 to -0.31] | -0.14 [-0.22 to -0.06]
  Rhinorrhea | -0.34 [-0.42 to -0.26] | -0.13 [-0.21 to -0.05]
  Nasal Congestion | -0.02 [-0.07 to 0.03] | 0.07 [0.03 to 0.12]
  Nasal Itching | -0.45 [-0.53 to -0.36] | -0.18 [-0.26 to -0.09]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Sneezing: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Sneezing was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.14]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Rhinorrhea: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Rhinorrhea was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.21, 95% CI 2-sided [-0.32 to -0.10]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Nasal Congestion: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Nasal Congestion was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p = 0.008, cLDA model; Difference in LS Means = -0.09, 95% CI 2-sided [-0.16 to -0.02]
Statistical Analysis 4: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Nasal Itching: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Nasal Itching was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.27, 95% CI 2-sided [-0.38 to -0.15]

6. Secondary Outcome: Change From Baseline to Week 2 in Each Nasal Symptom Sub-Score (Sneezing, Rhinorrhea, Nasal Congestion and Nasal Itching)
Description: Nasal symptoms sub-scores rated in the participant's diary included sneezing (daily frequency of attacks scored from 0 [<1 time or "none"] to 4 [≥21 times]), rhinorrhea (daily frequency of blowing nose scored from 0 [<1 time or "none"] to 4 [≥21 times]), nasal congestion (scored from 0 [no nasal blockage] to 4 [completely obstructed all day]), and nasal itching (scored from 0 [none] to 4 [nose is itchy, requiring frequent rubbing or blowing nose). Nasal symptom sub-scores ranged from 0 to 4, with a higher score indicating more frequent/severe nasal symptoms. BL measurement was an average of scores for 3 days prior to treatment (during Confirmation of Symptom Period). Post-BL measurement for Week 2 was an average of scores from Day 8 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 8 to 13 (Week 2 average) of double-blind treatment
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Sneezing | -0.51 [-0.60 to -0.42] | -0.27 [-0.35 to -0.18]
  Rhinorrhea | -0.49 [-0.58 to -0.40] | -0.24 [-0.33 to -0.16]
  Nasal Congestion | -0.03 [-0.09 to 0.03] | 0.06 [-0.00 to 0.12]
  Nasal Itching | -0.65 [-0.75 to -0.55] | -0.39 [-0.49 to -0.29]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Sneezing: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Sneezing was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.36 to -0.13]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Rhinorrhea: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Rhinorrhea was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.37 to -0.12]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Nasal Congestion: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Nasal Congestion was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p = 0.037, cLDA model; Difference in LS Means = -0.09, 95% CI 2-sided [-0.18 to -0.01]
Statistical Analysis 4: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Nasal Itching: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Nasal Itching was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.26, 95% CI 2-sided [-0.40 to -0.12]

7. Secondary Outcome: Change From Baseline in Each Nasal Symptom Sub-Score (Sneezing, Rhinorrhea, Nasal Congestion and Nasal Itching) During 2 Weeks of Therapy
Description: Nasal symptoms sub-scores rated in the participant's diary included sneezing (daily frequency of attacks scored from 0 [<1 time or "none"] to 4 [≥21 times]), rhinorrhea (daily frequency of blowing nose scored from 0 [<1 time or "none"] to 4 [≥21 times]), nasal congestion (scored from 0 [no nasal blockage] to 4 [completely obstructed all day]), and nasal itching (scored from 0 [none] to 4 [nose is itchy, requiring frequent rubbing or blowing nose). Nasal symptom sub-scores ranged from 0 to 4, with a higher score indicating more frequent/severe nasal symptoms. BL measurement was an average of scores for 3 days prior to treatment (during Confirmation of Symptom Period). Post-BL measurement for 2 week Average was an average of scores from Day 1 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to Day 13 (Weeks 1 through 2 average)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Sneezing | -0.44 [-0.52 to -0.37] | -0.20 [-0.27 to -0.12]
  Rhinorrhea | -0.41 [-0.48 to -0.33] | -0.18 [-0.26 to -0.11]
  Nasal Congestion | -0.02 [-0.07 to 0.03] | 0.07 [0.02 to 0.12]
  Nasal Itching | -0.54 [-0.62 to -0.46] | -0.27 [-0.36 to -0.19]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL in Sneezing During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Sneezing was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.14]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL in Rhinorrhea During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Rhinorrhea was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.23, 95% CI 2-sided [-0.33 to -0.12]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL in Nasal Congestion During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Nasal Congestion was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p = 0.009, cLDA model; Difference in LS Means = -0.09, 95% CI 2-sided [-0.16 to -0.02]
Statistical Analysis 4: Comparison: Desloratadine vs Placebo; Change from BL in Nasal Itching During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Nasal Itching was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value. cLDA model; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.26, 95% CI 2-sided [-0.38 to -0.15]

8. Secondary Outcome: Change From Baseline to Week 1 in Eye Symptoms (Pruritus, Watering Eyes and the Worse One of Either Pruritus or Watering Eyes)
Description: Eye symptoms rated in the participant's diary included eye pruritis (eye itching scored from 0 [none] to 4 [severe eye itching, requiring frequent rubbing of eye]) and watering eyes (scored from 0 [none] to 4 [severe eye watering requiring frequent wiping of eyes]). Eye symptom scores ranged from 0 to 4, with a higher score indicating greater severity of symptom. The change from baseline in eye pruritis, eye watering, and the worse one of either eye symptom were reported. Baseline measurement was an average of scores for 3 days prior to treatment. Post-baseline measurement for Week 1 was an average of scores from Day 1 to Day 7. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to 7 (Week 1 average) of double-blind treatment
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Eye Pruritus | -0.34 [-0.41 to -0.26] | -0.09 [-0.17 to -0.01]
  Watering Eyes | -0.17 [-0.24 to -0.11] | -0.02 [-0.08 to 0.05]
  Worse of Pruritus or Watering Eyes | -0.34 [-0.42 to -0.27] | -0.09 [-0.17 to -0.01]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Eye Pruritus: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Eye Pruritus was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.15]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Watering Eyes: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Watering Eyes was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.16, 95% CI 2-sided [-0.24 to -0.08]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Worse of Pruritus or Watering Eyes: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in the worse symptom of Pruritus or Watering Eyes estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.15]

9. Secondary Outcome: Change From Baseline to Week 2 in Eye Symptoms (Pruritus, Watering Eyes and the Worse One of Either Pruritus or Watering Eyes)
Description: Eye symptoms rated in the participant's diary included eye pruritis (eye itching scored from 0 [none] to 4 [severe eye itching, requiring frequent rubbing of eye]) and watering eyes (scored from 0 [none] to 4 [severe eye watering requiring frequent wiping of eyes]). Eye symptom scores ranged from 0 to 4, with a higher score indicating greater severity of symptom. The change from baseline in eye pruritis, eye watering, and the worse one of either eye symptom were reported. Baseline measurement was an average of scores for 3 days prior to treatment. Post-BL measurement for Week 2 was an average of scores from Day 8 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 8 to 13 (Week 2) of double-blind treatment
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Eye Pruritus | -0.56 [-0.66 to -0.46] | -0.32 [-0.41 to -0.22]
  Watering Eyes | -0.26 [-0.34 to -0.18] | -0.13 [-0.20 to -0.05]
  Worse of Pruritus or Watering Eyes | -0.56 [-0.66 to -0.46] | -0.32 [-0.41 to -0.22]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Eye Pruritus: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Eye Pruritus was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.37 to -0.12]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Watering Eyes: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Watering Eyes was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p = 0.010, cLDA model; Difference in LS Means = -0.13, 95% CI 2-sided [-0.24 to -0.03]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Worse of Pruritus or Watering Eyes: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in the worse symptom of Pruritus or Watering Eyes estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.24, 95% CI 2-sided [-0.37 to -0.12]

10. Secondary Outcome: Change From Baseline in Eye Symptoms (Pruritus, Watering Eyes and the Worse One of Either Pruritus or Watering Eyes) During 2 Weeks of Therapy
Description: Eye symptoms rated in the participant's diary included eye pruritis (eye itching scored from 0 [none] to 4 [severe eye itching, requiring frequent rubbing of eye]) and watering eyes (scored from 0 [none] to 4 [severe eye watering requiring frequent wiping of eyes]). Eye symptom scores ranged from 0 to 4, with a higher score indicating greater severity of symptom. The change from baseline in eye pruritis, eye watering, and the worse one of either eye symptom were reported. BL measurement was an average of scores for 3 days prior to treatment. Post-BL measurement for 2 week Average was an average of scores from Day 1 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to Day 13 (Weeks 1 through 2 average)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Eye Pruritus | -0.44 [-0.52 to -0.36] | -0.19 [-0.27 to -0.12]
  Watering Eyes | -0.21 [-0.27 to -0.15] | -0.07 [-0.13 to -0.00]
  Worse of Pruritus or Watering Eyes | -0.44 [-0.52 to -0.36] | -0.19 [-0.27 to -0.12]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL in Eye Pruritus During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Eye Pruritus was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.14]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL in Watering Eyes During 2 Weeks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Watering Eyes was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1 to Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.15, 95% CI 2-sided [-0.23 to -0.07]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; The LS mean change from BL to post BL (average score of 2 weeks) in the worse of Pruritus or Watering Eyes was estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1-Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.25, 95% CI 2-sided [-0.35 to -0.15]

11. Secondary Outcome: Change From Baseline in Interference With Daily Activities Score at Week 1, Week 2, and During 2 Weeks of Therapy
Description: Interference of allergic rhinitis symptoms with overall daily activities (such as work, study, housekeeping, sleep, or outing) was rated by the participant according to the following scale: 0=none, 1= symptoms cause few troubles, 2=symptoms cause intermediate problems between 1 and 3, 3=nasal symptoms cause painful and complicating daily life, or 4 = symptoms make daily activities impossible. Interference with daily activities scores ranged from 0 to 4 maximum, with a higher score indicating greater interference with daily activities. Baseline measurement was an average of scores for 3 days prior to treatment. Post-baseline measurement for Week 1 was an average of scores from Day 1 to Day 7. Post-BL measurement for Week 2 was an average of scores from Day 8 to Day 13. Post-BL measurement for 2 week Average was an average of scores from Day 1 to Day 13. Change from BL = Post BL measurement - BL measurement.
Time Frame: Baseline, Day 1 to 7 (Week 1 average), Day 8 to 13 (Week 2 average), Day 1 to Day 13 (Weeks 1 through 2 average) of double-blind treatment
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 223 | 225
units on a scale
  Week 1 | -0.23 [-0.29 to -0.16] | -0.07 [-0.14 to -0.01]
  Week 2 | -0.34 [-0.42 to -0.26] | -0.14 [-0.22 to -0.06]
  2 Week Average | -0.28 [-0.34 to -0.21] | -0.10 [-0.17 to -0.04]
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Change from BL to Week 1 in Interference with Daily Activities: Desloratadine vs. Placebo The LS mean change from BL to Week 1 post BL in Interference with Daily Activities was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 1) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.16, 95% CI 2-sided [-0.24 to -0.07]
Statistical Analysis 2: Comparison: Desloratadine vs Placebo; Change from BL to Week 2 in Interference with Daily Activities: Desloratadine vs. Placebo The LS mean change from BL to Week 2 post BL in Interference with Daily Activities was estimated using a cLDA model, where both BL and post-BL measurements (average score of 1 week prior to Week 2) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo was evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.19, 95% CI 2-sided [-0.30 to -0.09]
Statistical Analysis 3: Comparison: Desloratadine vs Placebo; Change from BL in Interference with Daily Activities During 2 Wks: Desloratadine vs. Placebo The LS mean change from BL to post BL (average score of 2 weeks) in Interference with Daily Activities estimated using a cLDA model, where both BL and post-BL measurements (average score from Day 1-Day 13) were included in the response variable. The treatment difference in terms of LS mean change from BL between desloratadine 5 mg and placebo evaluated with the 95% confidence interval and P-value; Test type: Superiority or Other; p < 0.001, cLDA model; Difference in LS Means = -0.17, 95% CI 2-sided [-0.26 to -0.08]

12. Secondary Outcome: Percentage of Participants With Impression Assessments of "Better" or "Much Better" as Assessed by the Investigator at Week 2
Description: The investigator assessed the participant's symptoms of allergic rhinitis and nasal findings at the end of the study (2 week visit or discontinuation visit) compared with those at the start of the study period (based on their recollection/memory of the participant's symptoms, no formal baseline assessment) and evaluated their impression of study drug on effect according to 6 grades: Much better, Better, Slightly better, Unchanged, Worse, or Unevaluable. The evaluation result and reason for judgment (if needed) was recorded in the participant's case report form. The investigator's impression was evaluated based on the symptoms for allergic rhinitis, nasal findings and participant's own impression at Week 2. The percentage of participants with assessments of "Better" and "Much better" graded by the investigator (Investigator's Impression Rate) was reported and analyzed using Odds Ratio analysis.
Time Frame: From Baseline to Week 2
Population: Participants in the FAS (all randomized participants who took ≥1 dose of study treatment) with available impression data.
Measure: Number; unit: percentage of participants
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 222 | 224
percentage of participants
  Much better | 2.3 | 3.1
  Better | 26.1 | 17.9
  Better + Much better Total | 28.4 | 21.0
  Less than better Total | 71.6 | 79.0
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Impression Rate as Assessed by Investigator: Desloratadine 5 mg/Placebo Odds Ratio Impression was evaluated using a logistic model with impression rate (percentage of assessments of "Better" + "Much better") as a response variable and treatment and severity as factors. Odds ratio was estimated and tested. A point estimate of >1 indicated that desloratadine 5mg was more effective than placebo; Test type: Superiority or Other; p = 0.071, Regression, Logistic; Odds Ratio (OR) = 1.492, 95% CI 2-sided [0.966 to 2.303]

13. Secondary Outcome: Percentage of Participants With Impression Assessments of "Better" or "Much Better" as Assessed Participants at Week 2
Description: The participant evaluated their symptoms of allergic rhinitis at the end of the study (2 week visit or discontinuation visit) compared with those at the start of the study period (based on their recollection/memory of their symptoms, no formal baseline assessment) and recorded in their Subject Allergy Diary their impression of study drug on effect according to 6 grades: Much better, Better, Slightly better, Unchanged, Worse, or Unevaluable. The percentage of participants with assessments of "Better" and "Much better" graded by the participant (Participant's Impression Rate) was reported and analyzed using Odds Ratio analysis.
Time Frame: From Baseline to Week 2
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Desloratadine | Placebo
Number analyzed (Participants) | 222 | 224
percentage of participants
  Much better | 5.9 | 4.9
  Better | 30.6 | 16.1
  Better + Much better Total | 36.5 | 21.1
  Less than better Total | 63.5 | 78.9
Statistical Analysis 1: Comparison: Desloratadine vs Placebo; Impression Rate as Assessed by Participant: Desloratadine 5 mg/Placebo Odds Ratio Impression was evaluated using a logistic model with impression rate (percentage of assessments of "Better" + "Much better") as a response variable and treatment and severity as factors. Odds ratio was estimated and tested. A point estimate of >1 indicated that desloratadine 5mg was more effective than placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.149, 95% CI 2-sided [1.408 to 3.280]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks (Up to 2 weeks after last dose of study drug)
Description: APaT; all participants who received ≥1 dose of study treatment. One participant randomized to Desloratadine was not treated due to withdrawn consent.
Arm/Group | Desloratadine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/223 | 0/225
Other Adverse Events (participants affected / at risk) | 0/223 | 0/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desloratadine (N=223) | Placebo (N=225)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.